CLINICAL TRIAL: NCT00531817
Title: A Randomized, Double-blind, Parallel-group Study to Evaluate the Safety and Efficacy of Tocilizumab (TCZ) Versus Placebo in Combination With Disease Modifying Antirheumatic Drugs (DMARDs) in Patients With Moderate to Severe Active Rheumatoid Arthritis (RA)
Brief Title: A Study of Tocilizumab in Combination With DMARDs in Patients With Moderate to Severe Rheumatoid Arthritis
Acronym: ROSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ML21136
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Results first posted 2010-08-04 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Tocilizumab 8 mg/kg + DMARDs (Experimental)
  Interventions: Drug: Tocilizumab; Drug: Permitted DMARDs
- Placebo + DMARDs (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Permitted DMARDs

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab intravenously at a dose of 8 mg/kg over a 1-hour infusion, every 4 weeks, for a total of 6 infusions.
  Other Names: Actemra; RoActemra
  Arms: Tocilizumab 8 mg/kg + DMARDs
Drug: Placebo — Placebo IV over a 1-hour infusion, every 4 weeks, for a total of 6 infusions.
  Arms: Placebo + DMARDs
Drug: Permitted DMARDs — As prescribed. The following DMARDs were permitted in this study: methotrexate (MTX), chloroquine, hydroxychloroquine, parenteral gold, sulfasalazine, azathioprine, and leflunomide. These DMARDs could be used alone or in combination, except for the combination of MTX and leflunomide, which was not allowed.

SUMMARY:
This 2-arm study assessed the safety and efficacy of tocilizumab versus placebo, both in combination with disease modifying antirheumatic drugs (DMARDs), in regard to reduction in signs and symptoms, in patients with moderate to severe active rheumatoid arthritis with an inadequate response to DMARDs. Patients were randomized in a ratio of 2:1 to receive either tocilizumab 8 mg/kg intravenously (IV) or placebo IV every 4 weeks. All patients also received stable antirheumatic therapy, including permitted DMARDs. The anticipated time on study treatment was 3-12 months and the target sample size was 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, ≥18 years of age
* Active rheumatoid arthritis of >6 months duration
* Received permitted DMARDs each at a stable dose for at least 7 weeks prior to baseline

Exclusion Criteria:

* Rheumatic autoimmune disease or inflammatory joint disease other than rheumatoid arthritis
* Major surgery within 8 weeks prior to screening or planned within 6 months following randomization
* Unsuccessful treatment with a biologic agent, including an anti-TNF agent
* Previous treatment with tocilizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 619 (Actual)
Dates: Start 2007-10; Primary Completion 2009-06 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (139):
- United States (138):
  - Birmingham, Alabama
  - Montgomery, Alabama
  - Lake Havasu City, Arizona
  - Paradise Valley, Arizona
  - Peoria, Arizona
  - Scottsdale, Arizona
  - Jonesboro, Arkansas
  - Beverly Hills, California
  - Escondido, California
  - La Jolla, California
  - Long Beach, California
  - Los Angeles, California
  - Pasadena, California
  - Santa Maria, California
  - Santa Monica, California
  - Upland, California
  - Van Nuys, California
  - Walnut Creek, California
  - Whittier, California
  - Colorado Springs, Colorado
  - Trumbull, Connecticut
  - Washington D.C., District of Columbia
  - Dunedin, Florida
  - Fort Lauderdale, Florida
  - Lake Mary, Florida
  - Melbourne, Florida
  - Miami, Florida
  - Ocala, Florida
  - Orange Park, Florida
  - Orlando, Florida
  - Palm Harbor, Florida
  - Plantation, Florida
  - Sarasota, Florida
  - Tamarac, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Blue Ridge, Georgia
  - Fort Valley, Georgia
  - Tifton, Georgia
  - Boise, Idaho
  - Idaho Falls, Idaho
  - Nampa, Idaho
  - Downers Grove, Illinois
  - Springfield, Illinois
  - Evansville, Indiana
  - Munster, Indiana
  - South Bend, Indiana
  - Leawood, Kansas
  - Bowling Green, Kentucky
  - Lexington, Kentucky
  - Baton Rouge, Louisiana
  - Monroe, Louisiana
  - New Orleans, Louisiana
  - Wheaton, Maryland
  - Mansfield, Massachusetts
  - Worcester, Massachusetts
  - Kalamazoo, Michigan
  - Saint Clair Shores, Michigan
  - Eagan, Minnesota
  - Flowood, Mississippi
  - Tupelo, Mississippi
  - Florissant, Missouri
  - St Louis, Missouri
  - Billings, Montana
  - Kalispell, Montana
  - Missoula, Montana
  - Grand Island, Nebraska
  - Las Vegas, Nevada
  - Reno, Nevada
  - Dover, New Hampshire
  - Freehold, New Jersey
  - New Brunswick, New Jersey
  - Passaic, New Jersey
  - Teaneck, New Jersey
  - Mineola, New York
  - New York, New York
  - Orchard Park, New York
  - Smithtown, New York
  - The Bronx, New York
  - Belmont, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Greensboro, North Carolina
  - Greenville, North Carolina
  - Hickory, North Carolina
  - Rock Hill, North Carolina
  - Akron, Ohio
  - Beechwood, Ohio
  - Mayfield, Ohio
  - Middleburg Heights, Ohio
  - Perrysburg, Ohio
  - Zanesville, Ohio
  - Norman, Oklahoma
  - Oklahoma City, Oklahoma
  - Lake Oswego, Oregon
  - Portland, Oregon
  - Salem, Oregon
  - Bethlehem, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Wexford, Pennsylvania
  - Willow Grove, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Florence, South Carolina
  - Greenville, South Carolina
  - Myrtle Beach, South Carolina
  - Rapid City, South Dakota
  - Sioux Falls, South Dakota
  - Watertown, South Dakota
  - Crossville, Tennessee
  - Hendersonville, Tennessee
  - Jackson, Tennessee
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Amarillo, Texas
  - Bellaire, Texas
  - Carrollton, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Mesquite, Texas
  - San Antonio, Texas
  - Temple, Texas
  - Waco, Texas
  - Salt Lake City, Utah
  - Burlington, Vermont
  - Burke, Virginia
  - Reston, Virginia
  - Salem, Virginia
  - Seattle, Washington
  - Spokane, Washington
  - Beckley, West Virginia
  - Clarksburg, West Virginia
  - Milwaukee, Wisconsin
  - Onalaska, Wisconsin
  - Wausau, Wisconsin
- San Juan, Puerto Rico

REFERENCES:
- [Derived] Yazici Y, Curtis JR, Ince A, Baraf HS, Lepley DM, Devenport JN, Kavanaugh A. Early effects of tocilizumab in the treatment of moderate to severe active rheumatoid arthritis: a one-week sub-study of a randomised controlled trial (Rapid Onset and Systemic Efficacy [ROSE] Study). Clin Exp Rheumatol. 2013 May-Jun;31(3):358-64. Epub 2013 Jan 10. PMID 23305631
- [Derived] Yazici Y, Curtis JR, Ince A, Baraf H, Malamet RL, Teng LL, Kavanaugh A. Efficacy of tocilizumab in patients with moderate to severe active rheumatoid arthritis and a previous inadequate response to disease-modifying antirheumatic drugs: the ROSE study. Ann Rheum Dis. 2012 Feb;71(2):198-205. doi: 10.1136/ard.2010.148700. Epub 2011 Sep 26. PMID 21949007

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab 8 mg/kg + DMARDs: Tocilizumab intravenously at a dose of 8 mg/kg over a 1-hour infusion, every 4 weeks, for a total of 6 infusions.
- Placebo + DMARDs: Placebo IV over a 1-hour infusion, every 4 weeks, for a total of 6 infusions.
Period: Randomized
Arm/Group | Tocilizumab 8 mg/kg + DMARDs | Placebo + DMARDs
Started | 412 | 207
Received Study Drug in Core Study | 409 (3 patients did not receive any study medication. Intent-to-treat population = 409.) | 205 (2 patients did not receive any study medication. Intent-to-treat population = 205.)
Completed | 353 | 173
Not Completed | 59 | 34
Period: Entered Extended Treatment Period
Arm/Group | Tocilizumab 8 mg/kg + DMARDs | Placebo + DMARDs
Started | 343 (Eligible patients completing core study could participate in extension at investigator's discretion.) | 170 (Eligible patients completing core study could participate in extension at investigator's discretion.)
Completed | 206 | 113
Not Completed | 137 | 57

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tocilizumab 8 mg/kg + DMARDs | Placebo + DMARDs | Total
Number analyzed (Participants) | 409 | 205 | 614
Age Continuous [Mean (Standard Deviation); unit: years] — Intent-to-treat population: Tocilizumab 8 mg/kg + DMARDs, n = 409 and Placebo + DMARDs, n = 205
  years | 55.2 (12.06) | 55.8 (12.42) | 55.5 (12.24)
Sex: Female, Male [Count of Participants; unit: Participants] — Intent-to-treat population: Tocilizumab 8 mg/kg + DMARDs, n = 409 and Placebo + DMARDs, n = 205
  Participants
    Female | 325 | 172 | 497
    Male | 84 | 33 | 117

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Patients With an Improvement of at Least 20%, 50%, or 70% in American College of Rheumatology (ACR) Score (ACR20, ACR50, ACR70) From Baseline at Weeks 4, 8, 12, 16, 20, and 24
Description: Improvement must be seen in tender and swollen joint counts and in at least 3 of the following 5 parameters. Patient and physician assessment of patient disease activity (DA) in previous 24 hours on a visual analog scale (VAS, no DA to maximum DA); patient assessment of pain in previous 24 hours on a VAS (none to unbearable); Health Assessment Questionnaire-Disability Index (20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities, 0=without difficulty to 3=unable to do); and C reactive protein or, if missing, erythrocyte sedimentation rate.
Time Frame: Baseline to Weeks 4, 8, 12, 16, 20, 24
Population: Intent-to-treat population: All randomized patients who received at least 1 dose of study medication. In determining ACR status, a last observation carried forward (LOCF) approach was used for missing joint count data. Patients with missing data or who escaped were classified as non-responders.
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab 8 mg/kg + DMARDs | Placebo + DMARDs
Number analyzed (Participants) | 409 | 205
Percentage of participants
  ACR20, Week 4 | 34.2 | 17.6
  ACR20, Week 8 | 46.5 | 25.4
  ACR20, Week 12 | 49.6 | 28.8
  ACR20, Week 16 | 47.7 | 28.8
  ACR20, Week 20 | 45.2 | 25.9
  ACR20, Week 24 | 44.7 | 25.4
  ACR50, Week 4 | 12.5 | 3.4
  ACR50, Week 8 | 20.8 | 5.4
  ACR50, Week 12 | 25.2 | 14.1
  ACR50, Week 16 | 26.7 | 15.1
  ACR50, Week 20 | 28.4 | 12.7
  ACR70, Week 4 | 4.4 | 1.5
  ACR70, Week 8 | 6.8 | 0.5
  ACR70, Week 12 | 11.5 | 4.9
  ACR70, Week 16 | 12.5 | 3.4
  ACR70, Week 20 | 16.9 | 5.4
  ACR70, Week 24 | 15.4 | 1.5

2. Primary Outcome: Percentage of Patients With an Improvement of at Least 50% in American College of Rheumatology (ACR) Score (ACR50) From Baseline at Week 24
Description: Improvement must be seen in tender and swollen joint counts and in at least 3 of the following 5 parameters. Patient and physician assessment of patient disease activity (DA) in previous 24 hours on a visual analog scale (VAS, no DA to maximum DA); patient assessment of pain in previous 24 hours on a VAS (none to unbearable); Health Assessment Questionnaire-Disability Index (20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities, 0=without difficulty to 3=unable to do); and C-reactive protein or, if missing, erythrocyte sedimentation rate.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab 8 mg/kg + DMARDs | Placebo + DMARDs
Number analyzed (Participants) | 409 | 205
Percentage of participants | 30.1 | 11.2
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg + DMARDs vs Placebo + DMARDs; Power calculation: Assuming placebo+DMARDs response rate of 15% and tocilizumab 8 mg/kg+DMARDs response rate of 28% based on previous trials, a sample size of 570 patients (2:1 ratio, tocilizumab+DMARDs n=380 and placebo+DMARDs n=190) will provide > 90% power to detect a difference between 2 treatment arms with 5% Type I error with a 2-sided Fisher's exact test. Null Hypothesis: The percentage of patients responding in each treatment group (tocilizumab+DMARDs vs placebo+ DMARDs) is the same; Test type: Superiority or Other; p < 0.0001, Fisher Exact — The p-value was not adjusted. The primary objective was a single comparison with an a priori threshold of 0.05 for statistical significance; Mean Difference (Final Values) = 18.85, 95% CI 2-sided [12.29 to 25.42]

3. Secondary Outcome: Mean Change From Baseline in Disease Activity Score 28 (DAS28) at Weeks 4, 8, 12, 16, 20, and 24
Description: DAS28 was calculated using the following formula: 0.56 × sqrt(TJC) + 0.28 × sqrt(SJC) + 0.70 × ln(ESR) + 0.014 × GH, where TJC = tender joint count on 28 joints, SJC = swollen joint count on 28 joints, ESR = erythrocyte sedimentation rate at the current visit (mm/hr), and GH = general health, ie, the patient's global assessment of disease activity (DA) in the previous 24 hours on a 100 mm visual analog scale (no DA to maximum DA). The DAS28 score ranges from 0 to 10, with higher scores indicating more rheumatoid arthritis. A negative change score indicates improvement.
Time Frame: Baseline to Weeks 4, 8, 12, 16, 20, 24
Population: Intent-to-treat population: All randomized patients who received at least 1 dose of study medication. No imputation of missing data was made; only observed data are reported.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab 8 mg/kg + DMARDs | Placebo + DMARDs
Number analyzed (Participants) | 409 | 205
Units on a scale
  Week 4, n=391, 194 | -1.77 (1.264) | -0.45 (1.065)
  Week 8, n= 382, 190 | -2.32 (1.454) | -0.72 (1.047)
  Week 12, n=361, 188 | -2.63 (1.433) | -0.97 (1.242)
  Week 16, n=343, 183 | -2.63 (1.605) | -0.93 (1.289)
  Week 20, n=273, 120 | -3.14 (1.535) | -1.36 (1.353)
  Week 24, n=265, 116 | -3.18 (1.526) | -1.23 (1.273)

4. Secondary Outcome: Percentage of Patients With European League Against Rheumatism (EULAR) Good, Moderate, or no Response at Weeks 4, 8, 12, 16, 20, and 24
Description: Change of the DAS28 score from baseline was used to determine the EULAR responses of good, moderate, or no response. For a post-baseline score ≤ 3.2, a change from baseline of < -1.2 was a good response, < -0.6 to ≥ -1.2 was a moderate response, and ≥ -0.6 was no response. For a post-baseline score > 3.2 to ≤ 5.1, a change from baseline of < -0.6 was a moderate response and ≥ -0.6 was no response. For a post-baseline score > 5.1, a change from baseline < -1.2 was a moderate response and ≥ -1.2 was no response. A good response could not be achieved for post-baseline scores > 3.2.
Time Frame: Baseline to Weeks 4, 8, 12, 16, 20, and 24
Population: Intent-to-treat population: All randomized patients who received at least 1 dose of study medication. Missing data was imputed as "no response".
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab 8 mg/kg + DMARDs | Placebo + DMARDs
Number analyzed (Participants) | 409 | 205
Percentage of participants
  Good response, Week 4 | 13.2 | 2.0
  Good response, Week 8 | 23.5 | 1.0
  Good response, Week 12 | 28.1 | 5.9
  Good response, Week 16 | 29.8 | 4.9
  Good response, Week 20 | 31.5 | 6.8
  Good response, Week 24 | 32.5 | 5.9
  Moderate response, Week 4 | 57.2 | 23.9
  Moderate response, Week 8 | 52.6 | 35.6
  Moderate response, Week 12 | 50.6 | 35.6
  Moderate response, Week 16 | 40.6 | 36.6
  Moderate response, Week 20 | 30.6 | 28.8
  Moderate response, Week 24 | 27.4 | 27.8
  No response, Week 4 | 29.6 | 74.1
  No response, Week 8 | 24.0 | 63.4
  No response, Week 12 | 21.3 | 58.5
  No response, Week 16 | 29.6 | 58.5
  No response, Week 20 | 37.9 | 64.4
  No response, Week 24 | 40.1 | 66.3

5. Secondary Outcome: Mean Change From Baseline in the Routine Assessment Patient Index Data (RAPID) Score at Weeks 4, 8, 12, 16, 20, and 24
Description: Derived from the Multidimensional Health Assessment Questionnaire (MDHAQ), the RAPID includes 3 domains that assess disease activity in rheumatoid arthritis: A physical function score (MDHAQ items 1a-j), a pain visual analog scale score (VAS, item 2 in the MDHAQ), and a global assessment of disease activity VAS score (item 6 in the MDHAQ). Each domain is scored on a scale of 0-10. The RAPID score is the sum of the 3 domain scores divided by 3 resulting in a total score on a scale of 0-10. Higher scores indicate more disease activity and a negative change from baseline indicates improvement.
Time Frame: Baseline to Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab 8 mg/kg + DMARDs | Placebo + DMARDs
Number analyzed (Participants) | 409 | 205
Units on a scale
  Week 4, n=403, 195 | -1.28 (1.921) | -0.50 (1.666)
  Week 8, n=392, 191 | -1.70 (2.087) | -0.73 (1.868)
  Week 12, n=379, 191 | -1.89 (2.244) | -0.99 (1.971)
  Week 16, n=358, 187 | -1.84 (2.286) | -0.86 (2.104)
  Week 20, n=292, 122 | -2.30 (2.212) | -1.51 (2.213)
  Week 24, n=283, 116 | -2.33 (2.294) | -1.29 (2.362)

6. Secondary Outcome: Mean Change From Baseline in 12-Item Short Form Health Survey v2 (SF-12) Scores at Weeks 4, 8, 12, 16, 20, and 24
Description: The SF-12 is a self-report measure of general health status with 1 or 2 items for each of 8 domains: Physical functioning, role limitations due to physical health problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health. Two component summaries, physical (PCS-12) and mental (MCS-12) were calculated using norm-based scoring, resulting in means of 50 and standard deviations of 10 in the 1998 general United States population. Higher scores represent better health and a positive change from baseline represents improvement.
Time Frame: Baseline to Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab 8 mg/kg + DMARDs | Placebo + DMARDs
Number analyzed (Participants) | 409 | 204
Units on a scale
  Physical component summary, Week 4, n=403, 197 | 4.14 (8.125) | 1.35 (7.501)
  Physical component summary, Week 8, n=393, 192 | 5.79 (8.862) | 1.95 (7.523)
  Physical component summary, Week 12, n=376, 192 | 7.17 (9.250) | 2.67 (8.098)
  Physical component summary, Week 16, n=358, 185 | 7.12 (9.278) | 2.40 (8.967)
  Physical component summary, Week 20, n=289, 123 | 8.43 (9.563) | 4.76 (8.855)
  Physical component summary, Week 24, n=283, 115 | 8.83 (9.931) | 3.57 (9.116)
  Mental component summary, Week 4, n=403, 197 | 2.91 (10.209) | 1.42 (9.379)
  Mental component summary, Week 8, n=393, 192 | 3.53 (10.719) | 2.18 (10.019)
  Mental component summary, Week 12, n=376, 192 | 3.29 (11.021) | 2.59 (10.848)
  Mental component summary, Week 16, n=358, 185 | 3.26 (10.845) | 2.23 (10.453)
  Mental component summary, Week 20, n=289, 123 | 4.33 (11.503) | 3.29 (10.760)
  Mental component summary, Week 24, n=283, 115 | 3.76 (12.284) | 3.39 (10.150)

7. Secondary Outcome: Mean Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Score at Weeks 4, 8, 12, 16, 20, and 24
Description: The FACIT-F is a 13-item patient self-report questionnaire that assesses fatigue over the previous 7 days by scoring each item on a 5-point scale (0=Not at all, 1=A little bit, 2=Somewhat, 3=Quite a bit, 4=Very much). An overall FACIT-F score was obtained by summing the scores of all 13 items. The overall score ranged from 0 to 52. A lower score indicates less fatigue. A negative change score indicates improvement.
Time Frame: Baseline to Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab 8 mg/kg + DMARDs | Placebo + DMARDs
Number analyzed (Participants) | 409 | 205
Units on a scale
  Week 4, n=405, 197 | 3.93 (8.786) | 3.06 (8.011)
  Week 8, n=394, 193 | 5.65 (10.039) | 3.85 (8.598)
  Week 12, n=378, 192 | 6.63 (10.504) | 3.91 (10.081)
  Week 16, n=358, 186 | 6.54 (10.876) | 3.62 (10.611)
  Week 20, n=289, 123 | 8.52 (11.147) | 6.24 (11.000)
  Week 24, n=283, 115 | 8.43 (11.513) | 5.89 (11.316)

8. Secondary Outcome: Mean Change From Baseline in the Medical Outcomes Study (MOS) Sleep Scale Score at Weeks 4, 8, 12, 16, 20, and 24
Description: The MOS Sleep Scale is a 12-item patient self-report instrument that assesses the quality and quantity of sleep over the previous 4 weeks. A sleep problems index (SLP9) was generated using 9 of the 12 items (1, 3, 4, 5, 6, 7, 8, 9, 12). Each item was normalized so that the lowest and highest possible scores were set to 0 and 100, respectively. The SLP9 score is the average of the recoded 9 items. The SLP9 score ranged from 0 to 100. Higher scores represent greater sleep problems. A negative change score indicates improvement.
Time Frame: Baseline to Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab 8 mg/kg + DMARDs | Placebo + DMARDs
Number analyzed (Participants) | 409 | 205
Units on a scale
  Week 4, n=405, 197 | -5.68 (14.334) | -3.87 (14.892)
  Week 8, n=394, 193 | -8.05 (14.384) | -6.77 (17.256)
  Week 12, n=378, 192 | -9.27 (16.824) | -4.80 (18.242)
  Week 16, n=358, 186 | -9.65 (17.117) | -5.42 (19.433)
  Week 20, n=291, 123 | 12.31 (17.991) | -10.89 (20.364)
  Week 24, n=283, 115 | -12.46 (19.167) | -10.11 (17.352)

9. Secondary Outcome: Mean Change From Baseline in Individual Components of the Routine Assessment Patient Index Data (RAPID) at Each Day During the First 7 Days of Treatment
Description: Derived from the Multidimensional Health Assessment Questionnaire (MDHAQ), the RAPID includes 3 domains that assess disease activity in rheumatoid arthritis: A physical function score (0-10), a pain visual analog scale score (VAS, 0-100), and a global assessment of disease activity VAS score (0-100). Each domain was assessed with the Patient Take Home Form (PTHF). Higher scores indicate more disease activity. A negative change score indicates improvement.
Time Frame: Baseline through Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab 8 mg/kg + DMARDs | Placebo + DMARDs
Number analyzed (Participants) | 409 | 205
Units on a scale
  Physical function, Day 1, n=372, 184 | -0.26 (1.203) | -0.22 (1.092)
  Physical function, Day 2, n=373, 183 | -0.35 (1.307) | -0.19 (1.197)
  Physical function, Day 3, n=370, 182 | -0.46 (1.376) | -0.09 (1.254)
  Physical function, Day 4, n=374, 184 | -0.50 (1.490) | -0.15 (1.342)
  Physical function, Day 5, n=372, 181 | -0.57 (1.499) | -0.27 (1.316)
  Physical function, Day 6, n=366, 179 | -0.65 (1.474) | -0.23 (1.356)
  Physical function, Day 7, n=354, 167 | -0.68 (1.518) | -0.33 (1.315)
  Pain VAS, Day 1, n=371, 183 | -10.50 (19.636) | -7.76 (18.498)
  Pain VAS, Day 2, n=373, 183 | -10.68 (21.439) | -8.79 (19.053)
  Pain VAS, Day 3, n=370, 182 | -12.60 (22.387) | -7.87 (21.506)
  Pain VAS, Day 4, n=374, 183 | -13.22 (23.202) | -8.46 (21.637)
  Pain VAS, Day 5, n=372, 179 | -13.53 (23.915) | -8.47 (21.536)
  Pain VAS, Day 6, n=366, 179 | -14.33 (24.608) | -7.98 (22.056)
  Pain VAS, Day 7, n=354, 166 | -14.68 (24.881) | -8.51 (21.148)
  Disease activity VAS, Day 1, n=372, 183 | -3.44 (19.690) | -1.32 (19.434)
  Disease activity VAS, Day 2, n=373, 183 | -3.87 (21.574) | -2.54 (19.562)
  Disease activity VAS, Day 3, n=370, 182 | -5.99 (22.090) | -2.19 (21.105)
  Disease activity VAS, Day 4, n=374, 183 | -5.72 (22.821) | -2.31 (21.131)
  Disease activity VAS, Day 5, n=371, 179 | -6.54 (23.256) | -2.93 (22.111)
  Disease activity VAS, Day 6, n=366, 179 | -7.90 (24.409) | -3.20 (21.936)
  Disease activity VAS, Day 7, n=354, 166 | -8.54 (23.836) | -3.50 (21.654)

10. Secondary Outcome: Percentage of Patients With an Improvement of at Least 20%, 50%, or 70% in American College of Rheumatology (ACR) Score (ACR20, ACR50, ACR70) From Baseline at Day 7
Description: as for outcome 1
Time Frame: Baseline to Day 7
Population: C-reactive protein (CRP) population: A subset of patients enrolled at designated study sites who met the CRP entry criteria (CRP ≥ 1 mg/dL), received at least 1 dose of study medication, and attended the Day 3 or Day 7 visit. LOCF was used for missing joint count data. Patients with missing data or who escaped were classified as non-responders.
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab 8 mg/kg + DMARDs | Placebo + DMARDs
Number analyzed (Participants) | 38 | 21
Percentage of participants
  ACR20 | 21 | 5
  ACR50 | 5 | 0
  ACR70 | 5 | 0

11. Secondary Outcome: Mean Change From Baseline in C-reactive Protein (CRP) at Days 3 and 7
Description: Serum concentration of CRP (high-sensitivity CRP [hsCRP] test) was analyzed by a central laboratory.
Time Frame: Baseline to Days 3 and 7
Population: C-reactive protein (CRP) population: A subset of patients enrolled at designated study sites who met the CRP entry criteria (CRP ≥ 1 mg/dL), received at least 1 dose of study medication, and attended the Day 3 or Day 7 visit. No imputation of missing data was made; only observed data are reported.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tocilizumab 8 mg/kg + DMARDs | Placebo + DMARDs
Number analyzed (Participants) | 40 | 22
mg/dL
  Day 3, n=38, 21 | -2.14 (2.391) | -0.52 (1.569)
  Day 7, n=38, 20 | -2.69 (2.854) | -0.31 (1.261)

ADVERSE EVENTS:
Time Frame: Adverse events that occurred in the double-blind treatment period and the extended treatment period are reported.
Description: Safety analysis population: All patients who received at least 1 dose of study medication and who had at least 1 post-baseline safety assessment. Placebo patients in the core study that received tocilizumab in the extension are reported in 2 groups resulting in a total of 787 patients in the 3 Adverse Events groups; only 619 enrolled in the study.
Groups:
- Tocilizumab + DMARDs: Initially treated with tocilizumab + DMARDs and received ≥ 1 dose of tocilizumab. The tocilizumab + DMARDs group includes all data (double-blind and extended treatment periods) for patients who were initially treated with tocilizumab in the double-blind treatment period. In the extended treatment period, patients received tocilizumab 8 mg/kg 1-hour IV infusion every 4 weeks (q4weeks) for up to 1 month post-commercial availability of tocilizumab in the United States.
- Placebo/Tocilizumab + DMARDs: Initially treated with placebo + DMARDs then received ≥ 1 dose of tocilizumab. The placebo/tocilizumab + DMARDs group includes all data collected after patients' first infusion of tocilizumab (whether escape therapy or extended treatment) for those who were initially treated with placebo in the double-blind treatment period. In the extended treatment period, patients received tocilizumab 8 mg/kg 1-hour IV infusion every 4 weeks (q4weeks) for up to 1 month post-commercial availability of tocilizumab in the United States.
- Placebo + DMARDs: Initially treated with placebo + DMARDs and received ≥ 1 dose of placebo. The placebo + DMARDs group includes all data collected while patients were on placebo for those who were initially treated with placebo in the double-blind treatment period.
Arm/Group | Tocilizumab + DMARDs | Placebo/Tocilizumab + DMARDs | Placebo + DMARDs
Serious Adverse Events (participants affected / at risk) | 79/409 | 27/173 | 11/205
Other Adverse Events (participants affected / at risk) | 259/409 | 98/173 | 69/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab + DMARDs (N=409) | Placebo/Tocilizumab + DMARDs (N=173) | Placebo + DMARDs (N=205)
Cellulitis (Infections and infestations) | 4 | 3 | 0
Pneumonia (Infections and infestations) | 8 | 3 | 0
Anal Abscess (Infections and infestations) | 1 | 0 | 0
Enterobacter Sepsis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis Viral (Infections and infestations) | 1 | 0 | 0
Lung Infection Pseudomonal (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 1 | 0
Septic Shock (Infections and infestations) | 1 | 0 | 0
Staphylococcal Infection (Infections and infestations) | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Diffuse Large B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1
Arteriosclerosis Coronary Artery (Cardiac disorders) | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 1
Coronary Artery Disease (Cardiac disorders) | 1 | 1 | 1
Myocardial Infarction (Cardiac disorders) | 2 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 3 | 3 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Jugular Vein Thrombosis (Vascular disorders) | 1 | 0 | 0
Haemorrhagic Stroke (Nervous system disorders) | 1 | 0 | 0
Loss of Consciousness (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 2 | 1 | 1
Chest Pain (General disorders) | 4 | 1 | 1
Biliary Dyskinesia (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 1 | 0 | 0
Calculus Ureteric (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Rash Vesicular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Swelling Face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Heart Rate Irregular (Investigations) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0
Bursitis infective staphylococcal (Infections and infestations) | 0 | 1 | 0
Cellulitis staphylococcal (Infections and infestations) | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Peptostreptococcus (Infections and infestations) | 0 | 1 | 0
Peridiverticular abscess (Infections and infestations) | 1 | 0 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 0 | 0
Pneumonia primary atypical (Infections and infestations) | 1 | 0 | 0
Puncture site infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Large cell carcinoma of the respiratory tract stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cardiovascular accident (Nervous system disorders) | 2 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
VIIIth nerve paralysis (Nervous system disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 3 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Aneurysm (Vascular disorders) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Drug abuse (Psychiatric disorders) | 0 | 1 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0
Skin graft (Surgical and medical procedures) | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab + DMARDs (N=409) | Placebo/Tocilizumab + DMARDs (N=173) | Placebo + DMARDs (N=205)
Upper Respiratory Tract Infection (Infections and infestations) | 70 | 28 | 10
Urinary Tract Infection (Infections and infestations) | 53 | 21 | 11
Diarrhoea (Gastrointestinal disorders) | 44 | 6 | 10
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 22 | 9 | 17
Sinusitis (Infections and infestations) | 44 | 17 | 5
Bronchitis (Infections and infestations) | 31 | 13 | 6
Nasopharyngitis (Infections and infestations) | 30 | 13 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 27 | 8 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 25 | 7 | 3
Nausea (Gastrointestinal disorders) | 25 | 9 | 5
Alanine aminotransferase increased (Investigations) | 31 | 9 | 3
Blood cholesterol increased (Investigations) | 23 | 6 | 0
Headache (Nervous system disorders) | 27 | 14 | 4
Hyperlipidaemia (Metabolism and nutrition disorders) | 25 | 13 | 3
Hypertension (Vascular disorders) | 23 | 9 | 1
Rash (Skin and subcutaneous tissue disorders) | 22 | 5 | 5
Fall (Injury, poisoning and procedural complications) | 20 | 10 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.